CLINICAL TRIAL: NCT03585257
Title: HEAL STUDY (Hepatic Encephalopathy and Albumin Study): A Double-Blind Randomized Controlled Trial Of Albumin In Hepatic Encephalopathy
Brief Title: HEAL STUDY (Hepatic Encephalopathy and Albumin Study)
Acronym: HEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: McGuire Research Institute (Other); Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAJAJ023
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cirrhosis; Hepatic Encephalopathy; Minimal Hepatic Encephalopathy; Covert Hepatic Encephalopathy
Keywords: covert hepatic encephalopathy; inflammation; cognition; quality of life
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Inflammation | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into receiving IV albumin vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV albumin (Experimental): 25% IV albutein (albumin) formulation will be infused 1.0g/kg IV over one hour weekly for 5 weeks
  Interventions: Biological: 25% IV albumin
- Placebo (Placebo Comparator): Normal saline will be infused 1.0g/kg IV over one hour weekly for 5 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 25% IV albumin — Intravenous 25% albumin infusion 1.0 g/kg body weight (maximum 100gm) once a week for five weeks for a maximum of 5 infusions. These infusions will be administered over sixty minutes per clinical treatment protocols for this population. Patients and investigators will be blinded as to the characteristic of the infusion. Pre-infusion serum albumin will be checked and if >4.0gm/dl, then normal saline will be given instead as mentioned in the blinding section above. Samples will be collected before and one hour after the infusion for all patients.
  The total grams of albumin infused over the 4 weeks during and outside the study will be collected and compared between groups.
  Arms: IV albumin
Other: Placebo — Normal saline infusion 1.0g/kg body weight once a week for five weeks for a maximum of 5 infusions. These infusions will be administered over sixty minutes per clinical treatment protocols for this population. Patients and investigators will be blinded as to the characteristic of the infusion. Pre-infusion serum albumin will be checked and if >4.0gm/dl, then normal saline will be given instead as mentioned in the blinding section above. Samples will be collected before and one hour after the infusion for all patients.
  The total grams of albumin infused over the 4 weeks during and outside the study will be collected and compared between groups.
  Arms: Placebo

SUMMARY:
Patients with continued cognitive impairment after episodes of HE have few options beyond lactulose and rifaximin in the US. Therefore using IV albumin in a randomized, double-blind, placebo-controlled trial, which could beneficially impact inflammation, could be an additional approach to improve cognition.

This 6 week trial will study changes in cognition, HRQOL and inflammation in patients with covert HE after prior overt HE using multiple IV albumin infusions vs. placebo.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a highly prevalent neuro-cognitive complication of cirrhosis characterized by cognitive dysfunction, and high rate of subsequent mortality and recurrence. HE also places a tremendous burden with a relentless increase in inpatient stay duration with charges topping $7244.7 million in 2009. There were almost 23,000 hospitalizations for HE in 2009 and far more patients with HE who are being managed as an outpatient in the US. In the NACSELD (North American Consortium for the Study of End-Stage Liver Disease) experience supported by Grifols, HE in inpatients is an independent risk factor for mortality and also the leading cause of readmissions in patients with cirrhosis.

HE has two major phases, an acute inpatient phase, where patients undergo evaluation for precipitating factors and HE treatment, and the post-discharge phase after HE resolution where the patient has a normal mental status but may be cognitively impaired. Furthermore, it is being increasingly recognized that even after the resolution of an acute HE episode with normal mental status and ability to understand and consent, patients do not regain their pre-HE cognitive function despite maximal therapy with the current standard of care. As many as 70% of patients with HE, despite standard of care, have residual significant cognitive impairments. Studies show that patients with HE, despite being on these medications which are standard of care, continue to have significant cognitive impairment translating into poor health-related quality of life (HRQOL), poor employment status, and very poor socio-economic status. This residual cognitive impairment is proportional to the number of HE episodes and places a heavy medical and socio-economic burden on patients, caregivers and society. In some cases, this approximates a dementia-like situation and makes this situation very difficult to manage.

These patients have three options in the current therapeutic situation which can improve brain function. However all of these options have problems in widespread acceptance or eligibility. First, if the patients are hyponatremic, correction of hyponatremia using tolvaptan can help but tolvaptan is now not FDA-approved for cirrhosis. Second a selected group of patients can undergo porto-systemic shunt embolization if their MELD score is <11 and they have a double shunt, which is the minority of individuals. Lastly a small trial done by our group showed improvement with fecal transplant but this requires several more years of study before this becomes mainstream.

Therefore, there is a major need for treating this continued cognitive impairment for which there are currently no widely-available therapeutic agents available but which can improve in selected cases. A medication or strategy that shows improvement in this functioning will be rapidly assimilated into the therapeutic algorithm and will potentially affect several thousand patients and their caregivers who continue to suffer from this issue.

There is strong evidence that this persistent cognitive impairment is accompanied by a sustained pro-inflammatory state that is not quenched by our current standard of care15. Ammonia, inflammation, endotoxemia, oxidative stress and endothelial dysfunction play an important role in the pathogenesis of HE. There is also evidence that in patients with advanced cirrhosis, i.e. those who are predisposed to HE, of reduction in albumin concentration and capacity to bind to these metabolites that precipitate HE.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Cirrhosis defined by any one of the following

   1. Cirrhosis on liver biopsy or transient wave elastography
   2. Nodular liver on imaging
   3. Endoscopic or radiological evidence of varices in a patient with chronic liver disease
   4. Platelet count <150,000/mm3 and AST/ALT ratio >1 in a patient with chronic liver disease
   5. Patients with frank decompensation (ascites, HE, variceal bleeding, hepato-pulmonary syndrome)
3. Prior HE controlled on standard of care therapy defined as lactulose or rifaximin for at least 2 months prior to enrollment.
4. Serum albumin <4 gm/dl
5. Cognitive impairment on any of the three testing strategies for HE including Psychometric hepatic encephalopathy score (PHES), Stroop test and Critical Flicker Frequency

   1. PHES aggregate score <-4SD based on norms published in Allampati et al located at the website www.encephalapp.com
   2. Stroop OffTime+OnTime values greater than norms published in Allampati et al located at the website www.encephalapp.com
   3. Critical Flicker Frequency value <39 Hz

Exclusion Criteria:

1. Unclear diagnosis of cirrhosis (does not meet the criteria outlined above)
2. No prior overt HE episodes
3. HE uncontrolled on standard of care defined as a mini-mental status exam<25
4. On regular IV albumin infusions due to scheduled paracentesis within the last 3 months
5. Recent alcohol abuse (within 3 months)
6. Unable to give consent
7. Current or recent invasive bacterial or fungal infections (<1 month)
8. Allergic reactions to IV albumin
9. Current or recent congestive heart failure (Systolic ejection fraction <25%) within the last year
10. Pregnancy (positive urine pregnancy test at screening)
11. In the opinion of the PI, those who are unlikely to survive 6 weeks or be able to adhere to the trial activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Improvement in psychometric hepatic encephalopathy score (PHES) from baseline vs end in albumin vs placebo group | 5 weeks
  Cognitive improvement on PHES
Minimal Hepatic Encephalopathy (MHE) reversal | 5 weeks
  change proportion of patients with MHE over time

SECONDARY OUTCOMES:
Change in SIckness Impact Profile (SIP) Questionnaire results from baseline vs end in albumin vs placebo group | 5 weeks
  Change in health-related quality of life
Change of PHES score to baseline in albumin group after discontinuation | 1 week
  Tracking PHES score after albumin discontinuation
Change of EncephalApp Stroop OffTime+OnTime to baseline in albumin group after discontinuation | 1 week
  Tracking Stroop score after albumin discontinuation
Change of CFF results to baseline in albumin group after discontinuation | 1 week
  Tracking CFF results after albumin discontinuation
Change of SIP score to baseline in albumin group after discontinuation | 1 week
  Tracking SIP results after albumin discontinuation
Change in EncephalApp Stroop OffTime+OnTime in seconds from baseline vs end in albumin vs placebo group | 5 weeks
  Change in EncephalApp Stroop
Change in Critical Flicker Frequency (CFF) results in Hz from baseline vs end in albumin vs placebo group | 5 weeks
  Change in CFF
Minimal hepatic encephalopathy(MHE) reversal to baseline in albumin group after discontinuation | 1 week
  relative proportion of patients in albumin who remained in MHE after albumin discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, MD, Principal Investigator — Hunter Holmes MVAMC
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fagan A, Gavis EA, Gallagher ML, Mousel T, Davis B, Puri P, Sterling RK, Luketic VA, Lee H, Matherly SC, Sanyal AJ, Stravitz RT, Patel V, Siddiqui MS, Asgharpour A, Fuchs M, Thacker L, Bajaj JS. A double-blind randomized placebo-controlled trial of albumin in outpatients with hepatic encephalopathy: HEAL study. J Hepatol. 2023 Feb;78(2):312-321. doi: 10.1016/j.jhep.2022.09.009. Epub 2022 Sep 22. PMID 36152764